CLINICAL TRIAL: NCT04376671
Title: Quantitative EEG Markers in Mild Cognitive Impairment in Epilepsy
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University 15
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Epilepsy
Keywords: Epilepsy, Mini Mental State Examination
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- temporal lobe epilepsy: Group of patients with temporal lobe epilepsy
  Interventions: Device: Electroencephalography
- Extra-temporal lobe epilepsy: Group of patients with extra-temporal lobe epilepsy
  Interventions: Device: Electroencephalography

INTERVENTIONS:
Device: Electroencephalography — The patients underwent EEG recordings according to previously published methods (Bonanni et al., 2008). . EEG recordings were analyzed with methods described in our previous work (Bonanni et al., 2008) by 2 experimenters unaware of the clinical conditions of the subjects. Briefly, quantitative EEGs (QEEGs) were recorded from 21 scalp derivations. Ag/AgCl disk scalp electrodes (19) were placed according to the international 10-20 system, EEG was recorded from Fp1, Fp2, Fz, F3, F4, F7, F8, Cz, C3, C4, Pz, P3, P4, T3, T 4, T5, T6, O1, and O2. Two additional electrodes were placed on A1 and A2. EEG activity was analyzed from single or multiple leads grouped to define the following scalp regions: anterior (Fz, Fp2, F7, Fp1, F3, F4, and F8), central (Cz, C3, and C4), posterior (Pz, P3, P4, O1, and O2), and temporal (T3, T4, T5, and T6).

SUMMARY:
Epileptic patients are plighted with limited daily activities, social dysfunction, family conflicts and cognitive impairment. Most of the studies had showed that cognitive disorders were frequent in patients with epilepsy.The cognitive impairment has been reported in around 25% of epileptic patients.

DETAILED DESCRIPTION:
Cognitive consequences in epilepsy are often described in the following domains: verbal memory, language, executive functions, and attention. However, most of the studies focus on one or two domains in a relatively small sample.

Few studies have investigated the influential factors for the epilepsy-related cognitive impairment . However, most of these studies merely focused on one or a few potential factors and failed to consider possible distractions from other influential factors. Therefore, it is crucial to include more potential factors in the analysis and to rule out possible confounding interactions between factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically confirmed epilepsy in adult patients.
* Non-symptomatic epilepsy.
* Normal CT or MRI brain, and
* Education level of primary school at least to respond to the scales correctly were included.

Exclusion Criteria:

* Psycho-neurological illnesses,
* History of alcoholism or drug abuse, or
* Recently on medications that may affect cognitive functions (like antidepressants and antipsychotic drugs).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 90 adult epileptic patients (according to the diagnosis of epilepsy in 2017, Fisher et al., 2017), 50 males and 40 females. With average age 24.5 ±5 .63.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Mini-mental state examination (MMSE) | 24 hours
  This is a rapid screening tool to estimate the cognitive functions that evaluates orientation, basic attention, working memory, learning, naming, construction, comprehension, and repetition. The maximum score is 30 and scores below 24 indicating cognitive impairment.
Montreal cognitive assessment (MoCA) | 24 hours
  Montreal cognitive assessment is a rapid sensitive screening tool for assessment of impaired cognitive function (Nasreddine et al., 2005). The main domains of MoCA scale include attention, executive functions, memory, language, attention, naming, orientation, and visual-spatial ability. The total score is 30 points. A score of 25 points or less indicated impaired cognitive function. For patients with less than12 years of education, one point was added to the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] England MJ, Liverman CT, Schultz AM, Strawbridge LM. Epilepsy across the spectrum: promoting health and understanding. A summary of the Institute of Medicine report. Epilepsy Behav. 2012 Oct;25(2):266-76. doi: 10.1016/j.yebeh.2012.06.016. Epub 2012 Oct 5. PMID 23041175
- [Background] Matonda-Ma-Nzuzi T, Mampunza Ma Miezi S, Mpembi MN, Mvumbi DM, Aloni MN, Malendakana F, Mpaka Mbeya D, Lelo GM, Charlier-Mikolajczak D. Factors associated with behavioral problems and cognitive impairment in children with epilepsy of Kinshasa, Democratic Republic of the Congo. Epilepsy Behav. 2018 Jan;78:78-83. doi: 10.1016/j.yebeh.2017.08.030. Epub 2017 Nov 25. PMID 29179103
- [Background] Bora E, Meletti S. Social cognition in temporal lobe epilepsy: A systematic review and meta-analysis. Epilepsy Behav. 2016 Jul;60:50-57. doi: 10.1016/j.yebeh.2016.04.024. Epub 2016 May 11. PMID 27179192
- [Background] Black LC, Schefft BK, Howe SR, Szaflarski JP, Yeh HS, Privitera MD. The effect of seizures on working memory and executive functioning performance. Epilepsy Behav. 2010 Mar;17(3):412-9. doi: 10.1016/j.yebeh.2010.01.006. Epub 2010 Feb 13. PMID 20153981
- [Background] Cassel A, Morris R, Koutroumanidis M, Kopelman M. Forgetting in temporal lobe epilepsy: When does it become accelerated? Cortex. 2016 May;78:70-84. doi: 10.1016/j.cortex.2016.02.005. Epub 2016 Feb 24. PMID 27010834
- [Background] Bonanni L, Thomas A, Tiraboschi P, Perfetti B, Varanese S, Onofrj M. EEG comparisons in early Alzheimer's disease, dementia with Lewy bodies and Parkinson's disease with dementia patients with a 2-year follow-up. Brain. 2008 Mar;131(Pt 3):690-705. doi: 10.1093/brain/awm322. Epub 2008 Jan 17. PMID 18202105
- [Derived] Elsherif M, Esmael A. Hippocampal atrophy and quantitative EEG markers in mild cognitive impairment in temporal lobe epilepsy versus extra-temporal lobe epilepsy. Neurol Sci. 2022 Mar;43(3):1975-1986. doi: 10.1007/s10072-021-05540-4. Epub 2021 Aug 18. PMID 34406537